CLINICAL TRIAL: NCT03395015
Title: Efficacia Del Trattamento Chirurgico Maxillo-facciale Sul Volto Dei Bambini Con Labiopalatoschisi: Valutazioni Estetiche ed Ortodontiche
Brief Title: Efficacy of Maxillo-facial Treatment on Cleft Lip and Palate Patients Faces: Aesthetic Considerations
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Prof. Massimo Cordaro (Unknown); Dr. Romeo Patini (Unknown); Dr. Oliva Giorgio (Unknown); Dr. Candida Ettore (Unknown); Dr. De Luca Marilisa (Unknown); Dr. Rizzo Maria Ida (Unknown); Dr. Zama Mario (Unknown); Dr. Rajabtork Zadeh Oriana (Unknown); Dr. Bucci Daria (Unknown); Prof. Gallenzi Patrizia (Unknown)
Responsible Party: Principal Investigator, Dr. Edoardo Staderini, PhD student, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 0027003/17
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Cleft Lip and Palate; Growth and Development; Cicatrix; Randomized Controlled Trial
Keywords: Reconstructive surgical procedures; Therapy, soft tissue; Treatment outcome; Outcome Assessment (Health Care); Photogrammetry; Physical Appearance, Body
MeSH Terms: conditions — Cleft Lip; Cicatrix

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Full-face 3-D images: 3-D images acquisition of CLP patients' faces at rest is set at different timepoints: 1 week preoperative, 1- and 6-months postoperative. Therefore, laypeople's assessment of the facial appearance of CLP patients is based on full facial views.
  Interventions: Other: VAS scale (from 1 to 10) esthetic assessment of facial 3-D images
- Nasolabial 3-D images: The control group is composed of cropped 3-D images of CLP patients' faces at rest, which show isolated nasolabial regions of CLP patients. The judgement of these pictures warrants an assessment based solely on the nasolabial appearance.
  Interventions: Other: VAS scale (from 1 to 10) esthetic assessment of facial 3-D images

INTERVENTIONS:
Other: VAS scale (from 1 to 10) esthetic assessment of facial 3-D images — The rating process is biphasic: firstly a 3-D model is showed to the raters, who can orientate the vultus, familiarize with the 3-D technology and have a first glance evaluation. Secondly, the judges are asked to rate each of the following patient views: right profile, left profile, frontal, neck hyperextension and hyperflexion views Two weeks after the first assessment, the same judges assessed the same number of pictures, once again in random order.

SUMMARY:
The aim of the study is to analyze the esthetic outcome of the first surgical repair of cleft lip and palate (CLP) patients.

The aim of the study is to identify differences in the aesthetic evaluation of full-face and nasolabial region 3-D images of CLP patients following primary lip repair by laypeople.

DETAILED DESCRIPTION:
The management of cleft lip and palate patient's generally involves the soft palate reconstruction as well as the repair of lip and nasal soft tissue defects.

From an esthetic point of view, the primary repair, usually performed between 9 and 18 months of age, prepares the patients to grow into childhood and succeed in life without focusing on their deformity.

An increasing number of outcome measure rating systems has been raised, suggesting a lack of consensus to a reliable, validated and reproducible scoring system for facial aesthetics in cleft patients. Many templates and lay panel scoring systems have been described, yet never fully validated. Advanced 3D imaging technologies may produce validated outcome measures in the future, but presently there remains a need to develop a robust method of facial aesthetic evaluation based on standardised patient photographs.

The aim of the study is to to determine and compare the level of agreement among examiners' subjective aesthetic evaluation of full-face and nasolabial region 3-D images of CLP patients following primary lip repair by laypeople, developing some recommendations for a consistent scoring protocol.

ELIGIBILITY:
Inclusion Criteria:

* age, between 20 and 25 years
* sex, in order to have at least 25 male and female raters
* sociocultural status: the layperson panel includes undergraduate students without extensive professional knowledge on cleft lip and palate patients

Exclusion Criteria:

* previous participation in research studies
* familiarity or close friendship with cleft lip and palate patients
* lack of blindness about the study protocol (it could bias the reported results)

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The raters selection is aiming to have an equal number of male and female judges.
Study Population: The lay panel consisted of 50 undergraduate students who had little or no training in cleft palate or cranio-facial treatment. All panelists were recruited from the Catholic University of Sacred Heart. The participation of the study is voluntary. A preliminary assessment of raters' knowledge has been performed through an oral examination.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Intrarater and interrater consistency | 3-D images are assessed twice, the timespan between the two evaluations is two weeks
  The primary outcome of this study is to compare intrarater and interrater reliability of the ratings in both groups.
  The reliability of a panel of 3 and 6 judges for the different scoreswere estimated by using the Cronbach alfa formula.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Cordaro, Medicine, Principal Investigator — Catholic University of the Sacred Hearth - Rome
Locations (1):
- Catholic University of the Sacred Heart, Roma, Italia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF
Time Frame: The data will be available as soon as the study will be registered. The informed consent form is written in italian

REFERENCES:
- [Result] Iliopoulos C, Mitsimponas K, Lazaridou D, Neukam FW, Stelzle F. A retrospective evaluation of the aesthetics of the nasolabial complex after unilateral cleft lip repair using the Tennison-Randall technique: a study of 44 cases treated in a single cleft center. J Craniomaxillofac Surg. 2014 Dec;42(8):1679-83. doi: 10.1016/j.jcms.2014.05.013. Epub 2014 May 24. PMID 24962045
- [Result] Eichenberger M, Staudt CB, Pandis N, Gnoinski W, Eliades T. Facial attractiveness of patients with unilateral cleft lip and palate and of controls assessed by laypersons and professionals. Eur J Orthod. 2014 Jun;36(3):284-9. doi: 10.1093/ejo/cjt047. Epub 2013 Jul 5. PMID 23832974
- [Result] de Ladeira PR, Alonso N. Protocols in cleft lip and palate treatment: systematic review. Plast Surg Int. 2012;2012:562892. doi: 10.1155/2012/562892. Epub 2012 Nov 1. PMID 23213503
- [Result] Sharma VP, Bella H, Cadier MM, Pigott RW, Goodacre TE, Richard BM. Outcomes in facial aesthetics in cleft lip and palate surgery: a systematic review. J Plast Reconstr Aesthet Surg. 2012 Sep;65(9):1233-45. doi: 10.1016/j.bjps.2012.04.001. Epub 2012 May 15. PMID 22591614
- [Result] Stebel A, Desmedt D, Bronkhorst E, Kuijpers MA, Fudalej PS. Rating nasolabial appearance on three-dimensional images in cleft lip and palate: a comparison with standard photographs. Eur J Orthod. 2016 Apr;38(2):197-201. doi: 10.1093/ejo/cjv024. Epub 2015 Apr 21. PMID 25900054
- [Result] Mosmuller DG, Bijnen CL, Kramer GJ, Disse MA, Prahl C, Kuik DJ, Niessen FB, Don Griot JP. The Asher-McDade Aesthetic Index in Comparison With Two Scoring Systems in Nonsyndromic Complete Unilateral Cleft Lip and Palate Patients. J Craniofac Surg. 2015 Jun;26(4):1242-5. doi: 10.1097/SCS.0000000000001784. PMID 26080166